CLINICAL TRIAL: NCT01839188
Title: A Phase 3 Open-label Study to Evaluate the Immunogenicity and Safety of a Mixed (HEXA/PENTA/HEXA) Primary Series Schedule That Includes V419 (PR5I) at 2 and 6 Months of Age and Pediacel at 4 Months of Age.
Brief Title: Spanish Mixed HEXA/PENTA/HEXA Schedule (V419-010)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MCM Vaccines B.V. (Industry)
Collaborators: Sanofi Pasteur, a Sanofi Company (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V419-010; 2012-004221-25 (EudraCT Number); PRI02C (Other: MCMVaccBV Protocol ID); V419-010 (Other: Merck Protocol Number)
Record Dates: First submitted 2013-04-19; First posted 2013-04-24 (Estimated); Results first posted 2019-02-25 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Neisseria Meningitidis; Bacterial Infections; Virus Diseases
MeSH Terms: conditions — Bacterial Infections; Virus Diseases | interventions — Vaxelis; diphtheria-tetanus-five component acellular pertussis-inactivated poliomyelitis -Haemophilus influenzae type b conjugate vaccine; RotaTeq; 13-valent pneumococcal vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PR5I (V1); Pediacel® (V2); PR5I (V3) (Experimental): [Vaccination 1]: Single doses of PR5I (V419) + NeisVac-C® + Prevenar 13® by intramuscular (IM) injection + oral RotaTeq®, given at 2 months of age. [Vaccination 2]: Single doses of Pediacel® + NeisVac-C® + Prevenar 13® by IM injection + oral RotaTeq®, given at 4 months of age. [Vaccination 3]: Single dose of PR5I (V419) by IM injection + oral RotaTeq®, given at 6 months of age.
  Interventions: Biological: PR5I; Biological: Pediacel®; Biological: NeisVac-C®; Biological: RotaTeq®; Biological: Prevenar 13®

INTERVENTIONS:
Biological: PR5I — Hexavalent PR5I vaccine (DTaP-HB-IPV-Hib = Diphtheria and Tetanus Toxoids and Acellular Pertussis Adsorbed [DTaP], Hepatitis B [HB; Recombinant DNA], Inactivated Poliovirus [IPV], and Haemophilus influenzae type b [Hib] conjugate vaccine [adsorbed]) at 0.5 mL for IM injection (left upper thigh) at 2 and 6 months of age.
  Other Names: V419; Vaxelis®; DTaP-HB-IPV-Hib
Biological: Pediacel® — Pentavalent Pediacel® vaccine (DTaP-IPV-Hib = Diphtheria and Tetanus Toxoids and Acellular Pertussis Adsorbed [DTaP], Inactivated Poliovirus [IPV], and Haemophilus influenzae type b [Hib] conjugate vaccine [adsorbed]) at 0.5 mL for IM injection (left upper thigh) at 4 months of age.
  Other Names: DTaP-IPV-Hib
Biological: NeisVac-C® — Meningococcal group C (MCC) polysaccharide conjugate vaccine (adsorbed) at 0.5 mL for IM injection (right upper thigh) at 2 and 4 months of age.
Biological: RotaTeq® — Human-bovine rotavirus reassortants (live) vaccine 2 mL oral administration at 2, 4 and 6 months of age. RotaTeq® administered prior to any other vaccine administration to avoid having the infant participants spit up the RotaTeq® when crying.
Biological: Prevenar 13® — Pneumococcal polysaccharide conjugate vaccine [PCV; 13-valent, adsorbed]) at 0.5 mL for IM injection (right upper thigh) at 2 and 4 months of age.
  Other Names: PCV-13

SUMMARY:
To evaluate the immune response and the safety of a primary series schedule that includes V419 (PR5I) at 2 and 6 months of age and Pediacel at 4 months of age

Primary objectives

* To demonstrate that the mixed schedule induces acceptable responses for Hepatitis B (HB) one month after completion of the mixed schedule
* To demonstrate that the mixed schedule induces acceptable responses for Haemophilus influenzae type b (Hib) one month after completion of the mixed schedule

Secondary objectives

* To describe the antibody response to all PR5I antigens one month after completion of the mixed schedule
* To describe the antibody response to meningococcal serogroup C (MCC) conjugate vaccine one month after the second dose of MenC vaccine
* To describe the safety profile after each dose of study vaccines administered

ELIGIBILITY:
Inclusion Criteria:

* Healthy infant 46 to 74 days (both inclusive)
* Documented receipt of only one dose of monovalent hepatitis B vaccine within the 3 days after birth
* Parent(s)/legal representative able to comply with the study procedures

Exclusion Criteria:

* Participation in any study with an investigational compound or device since birth
* History of congenital or acquired immunodeficiency
* Chronic illness that could interfere with study conduct or completion
* Hypersensitivity to any of the study vaccines components or history of a life-threatening reaction to a vaccine containing the same substances as the study vaccines
* Contraindication to Pediacel®, NeisVac-C®, Prevenar 13®, and RotaTeq®
* History or maternal history of HBsAg seropositivity
* Coagulation disorder that contraindicate intramuscular injection
* History of vaccination with a Haemophilus influenzae type b conjugate, diphtheria, tetanus, pertussis (acelullar or whole-cell), poliovirus, meningococcal serogroup C conjugate, pneumococcal conjugate containing vaccine(s)
* History of hepatitis B, Haemophilus influenzae type b, diphtheria, tetanus, pertussis, poliomyelitis, or serogroup C meningococcal infection
* Receipt of immune globulin, blood or blood-derived products since birth
* Receipt of systemic corticosteroids for more than 14 consecutive days within one month of the study start
* Identified as a natural or adopted child of the Investigator or employee with direct involvement in the proposed study

Ages: 46 Days to 76 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 385 (Actual)
Dates: Start 2013-05-01 (Actual); Primary Completion 2014-03-19 (Actual); Study Completion 2014-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Martinon-Torres F, Boisnard F, Thomas S, Sadorge C, Borrow R; PRI02C study group. Immunogenicity and safety of a new hexavalent vaccine (DTaP5-IPV-HB-Hib) administered in a mixed primary series schedule with a pentavalent vaccine (DTaP5-IPV-Hib). Vaccine. 2017 Jun 27;35(30):3764-3772. doi: 10.1016/j.vaccine.2017.05.043. Epub 2017 Jun 2. PMID 28583305

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled N=385 infant participants previously vaccinated with only 1 dose of monovalent Hepatitis B vaccine, within 3 days after birth, outside of study context.
Pre-assignment Details: Participants progressed through the study as a single group, with all participants receiving the same mixed-schedule vaccination series. Vaccination (V1) was administered on Study Day 0 (2 months of age), with V2 (4 months of age) and V3 (6 months of age) administered at Study Months 2 and 4, respectively.
Period: Overall Study
Arm/Group | PR5I (V1); Pediacel® (V2); PR5I (V3)
Started | 385
Treated | 385
Completed | 384 (N=1 treated participant withdrew before receiving V3)
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: All participants receiving ≥1 dose of study vaccination.
Arm/Group | PR5I (V1); Pediacel® (V2); PR5I (V3)
Number analyzed (Participants) | 385
Age, Continuous [Mean (Standard Deviation); unit: Days] | 60.72 (7.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 199
  Male | 186
Body Weight [Mean (Standard Deviation); unit: kg] — Population: Includes all participants receiving ≥1 dose of study vaccination, having available data for body weight.
  kg
    number analyzed (Participants) | 384
    (all) | 5.14 (0.59)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Anti-Hepatitis B Surface Antigen (HBsAg) Antibody Titer ≥10 mIU/mL
Description: The percentage of participants with an anti-HBsAg antibody titer ≥10 mill-International Units/mL (mIU/mL) was assessed. Participant serum samples were collected for analysis with an enhanced chemiluminescence assay to determine the concentration of antibodies to HBsAg.
Time Frame: Month 5 (one month after receiving Vaccination 3)
Population: All participants receiving ≥1 dose of study vaccination without protocol deviation, having post-vaccination immunogenicity data available for the evaluation of the respective analysis endpoint.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | PR5I (V1); Pediacel® (V2); PR5I (V3)
Number analyzed (Participants) | 369
Percentage of Participants | 98.9 [97.2 to 99.7]

2. Primary Outcome: Percentage of Participants With an Anti-Polyribosylribitol Phosphate (PRP) Antibody Titer ≥0.15 µg/mL
Description: The percentage of participants with an anti-Polyribosylribitol Phosphate (PRP) antibody titer ≥0.15 µg/mL was assessed. Participant serum samples were collected for analysis by radioimmunoassay to determine the concentration of antibodies to PRP, a Haemophilus influenzae type b (Hib) capsular polysaccharide.
Time Frame: Month 5 (one month after receiving Vaccination 3)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | PR5I (V1); Pediacel® (V2); PR5I (V3)
Number analyzed (Participants) | 365
Percentage of Participants | 100.0 [99.0 to 100.0]

3. Secondary Outcome: Geometric Mean Concentration of Antibodies to Hepatitis B Surface Antigen (HBsAg)
Description: Participant serum samples were collected for analysis with an enhanced chemiluminescence assay to determine the geometric mean concentration of antibodies to Hepatitis B Surface Antigen (HBsAg). The unit of measure is milli International Units/mL (mIU/mL).
Time Frame: Month 5 (one month after receiving Vaccination 3)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | PR5I (V1); Pediacel® (V2); PR5I (V3)
Number analyzed (Participants) | 369
mIU/mL | 1054.97 [911.49 to 1221.03]

4. Secondary Outcome: Geometric Mean Concentration of Antibodies to Polyribosylribitol Phosphate (PRP) Antigen
Description: Participant serum samples were collected for analysis by radioimmunoassay (RIA) to determine the geometric mean concentration of antibodies to polyribosylribitol phosphate (PRP), a Haemophilus influenzae type b (Hib) capsular polysaccharide.
Time Frame: Month 5 (one month after receiving Vaccination 3)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | PR5I (V1); Pediacel® (V2); PR5I (V3)
Number analyzed (Participants) | 365
μg/mL | 8.00 [7.17 to 8.93]

5. Secondary Outcome: Geometric Mean Concentration of Antibodies to Diphtheria Toxin
Description: Participant serum samples were collected for analysis with a Micrometabolic Inhibition Test (MIT) to determine the geometric mean concentration of neutralizing antibodies to diphtheria toxin. The unit of measure is International Units/mL (IU/mL).
Time Frame: Month 5 (one month after receiving Vaccination 3)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | PR5I (V1); Pediacel® (V2); PR5I (V3)
Number analyzed (Participants) | 359
IU/mL | 0.47 [0.42 to 0.52]

6. Secondary Outcome: Geometric Mean Concentration of Antibodies to Tetanus Toxin
Description: Participant serum samples were collected for analysis by Enzyme-linked Immunosorbent Assay (ELISA) to determine the geometric mean concentration of antibodies to tetanus toxin. The unit of measure is International Units/mL (IU/mL).
Time Frame: Month 5 (one month after receiving Vaccination 3)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | PR5I (V1); Pediacel® (V2); PR5I (V3)
Number analyzed (Participants) | 350
IU/mL | 2.44 [2.31 to 2.59]

7. Secondary Outcome: Geometric Mean Concentrations of Antibodies to Pertussis Antigens
Description: Participant serum samples were collected for analysis by ELISA to determine the geometric mean concentration of antibodies (Abs) to the following Pertussis antigens: pertussis toxoid (PT), filamentous hemagglutinin (FHA), pertactin (PRN) and fimbriae types (FIM) 2&3. The unit of measure is ELISA Units/mL (EU/mL).
Time Frame: Month 5 (one month after receiving Vaccination 3)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | PR5I (V1); Pediacel® (V2); PR5I (V3)
Number analyzed (Participants) | 349
EU/mL
  Anti-PT Abs | 107.46 [101.55 to 113.71]
  Anti-FHA Abs | 67.09 [62.38 to 72.15]
  Anti-PRN Abs | 56.46 [51.60 to 61.78]
  Anti-FIM 2&3 Abs | 360.99 [332.58 to 391.82]

8. Secondary Outcome: Geometric Mean Titers for Antibodies to Inactivated Poliovirus 1-3 (IPV1-3)
Description: Participant serum samples were collected for analysis with a Micrometabolic Inhibition Test (MIT) to determine the geometric mean titer of neutralizing antibodies (Abs) to Inactivated Poliovirus 1, 2, & 3 (IPV1, IPV2, & IPV3). The unit of measure is titer, expressed as the reciprocal dilution of the highest dilution that neutralizes 50% of the challenge virus.
Time Frame: Month 5 (one month after receiving Vaccination 3)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | PR5I (V1); Pediacel® (V2); PR5I (V3)
Number analyzed (Participants) | 356
Titer
  Anti-IPV1 Abs | 663.97 [588.10 to 749.62]
  Anti-IPV2 Abs | 1198.93 [1051.90 to 1366.51]
  Anti-IPV3 Abs | 764.64 [664.70 to 879.61]

9. Secondary Outcome: Percentage of Participants Responding to Polyribosylribitol Phosphate (PRP) Antigen, Diptheria Toxin (D), Tetanus Toxin (T), and Inactivated Poliovirus 1, 2, & 3 (IPV1, IPV2, & IPV3)
Description: Participants were considered as responding if the observed concentration or titer for antibodies (Abs) to specific antigens exceeded the following thresholds:
  1. For anti-PRP Abs (Hib capsular polysaccharide) - Response defined as a concentration ≥1 µg/mL (measured by RIA);
  2. For anti-D Abs - Response defined at 2 concentrations: ≥0.01 IU/mL and ≥0.10 IU/mL (measured by MIT);
  3. For anti-T Abs - Response defined at 2 concentrations: ≥0.01 IU/mL and ≥0.10 IU/mL (measured by ELISA);
  4. For anti-IPV1, anti-IPV2, and anti-IPV3 Abs - Response defined as a titer ≥ 8 (measured by MIT).
  The percentage of participants considered as responding to the individual antigen (per the response threshold[s]) were assessed.
Time Frame: Month 5 (one month after receiving Vaccination 3)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | PR5I (V1); Pediacel® (V2); PR5I (V3)
Number analyzed (Participants) | 370
Percentage of Participants
  Anti-PRP Ab ≥ 1 μg/mL: number analyzed (Participants) | 365
  Anti-PRP Ab ≥ 1 μg/mL | 95.3 [92.6 to 97.3]
  Anti-Diptheria Ab ≥0.01 IU/mL: number analyzed (Participants) | 359
  Anti-Diptheria Ab ≥0.01 IU/mL | 100.0 [99.0 to 100.0]
  Anti-Diptheria Ab ≥0.10 IU/mL: number analyzed (Participants) | 359
  Anti-Diptheria Ab ≥0.10 IU/mL | 92.2 [88.9 to 94.8]
  Anti-Tetanus ≥0.01 IU/mL: number analyzed (Participants) | 350
  Anti-Tetanus ≥0.01 IU/mL | 100.0 [99.0 to 100.0]
  Anti-Tetanus Ab ≥0.10 IU/mL: number analyzed (Participants) | 350
  Anti-Tetanus Ab ≥0.10 IU/mL | 100.0 [99.0 to 100.0]
  Anti-IPV1 Ab Titer ≥8: number analyzed (Participants) | 356
  Anti-IPV1 Ab Titer ≥8 | 100.0 [99.0 to 100.0]
  Anti-IPV2 Ab Titer ≥8: number analyzed (Participants) | 356
  Anti-IPV2 Ab Titer ≥8 | 100.0 [99.0 to 100.0]
  Anti-IPV3 Ab Titer ≥8: number analyzed (Participants) | 356
  Anti-IPV3 Ab Titer ≥8 | 100.0 [99.0 to 100.0]

10. Secondary Outcome: Geometric Mean Titer of Anti-Meningococcal Group C Polysaccharide Conjugate (MCC) Antibodies
Description: Participant serum samples were collected to determine the geometric mean titer of anti-MCC antibodies, measured by the Serum Bactericidal Antibody assay using rabbit complement (rSBA). The unit of measure is titer, expressed as the reciprocal of the final serum dilution giving ≥50% killing of the challenge bacterial strain.
Time Frame: Month 3 (one month after receiving Vaccination 2)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | PR5I (V1); Pediacel® (V2); PR5I (V3)
Number analyzed (Participants) | 375
Titer | 739.63 [659.94 to 828.96]

11. Secondary Outcome: Percentage of Participants With an Anti-Meningococcal Group C Polysaccharide Conjugate (MCC) Antibody Titer ≥8
Description: The percentage of participants with an anti-MCC antibody titer ≥8 was assessed. Participant serum samples were collected and analyzed for anti-MCC antibodies with the Serum Bactericidal Antibody assay using rabbit complement (rSBA).
Time Frame: Month 3 (one month after receiving Vaccination 2)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | PR5I (V1); Pediacel® (V2); PR5I (V3)
Number analyzed (Participants) | 375
Percentage of Participants | 99.2 [97.7 to 99.8]

12. Secondary Outcome: Percentage of Participants With a Body Temperature ≥38°C After Each Vaccination
Description: The percentage of participants with a body temperature ≥38.0°C from Day 1 to Day 5 after each vaccination was assessed. Per protocol, the participant's parent(s)/legal representative recorded daily body temperature measurements each evening by the axillary route (N=3 collected via rectal route; N=1 collected via oral route) and recorded these observations on the Vaccine Report Card (VRC). Temperatures were based on actual temperatures recorded with no adjustments for the route of assessment.
Time Frame: Up to Day 5 following each vaccination
Population: All participants receiving ≥1 dose of any vaccination with corresponding safety follow-up data, having available body temperature data.
Measure: Number; unit: Percentage of Participants
Groups:
- PR5I (V1): [Vaccination 1]: Single doses of PR5I (V419) + NeisVac-C® + Prevenar 13® by IM injection + oral RotaTeq®, given at 2 months of age.
- Pediacel® (V2): [Vaccination 2]: Single doses of Pediacel® + NeisVac-C® + Prevenar 13® by IM injection + oral RotaTeq®, given at 4 months of age.
- PR5I (V3): [Vaccination 3]: Single dose of PR5I (V419) by IM injection + oral RotaTeq®, given at 6 months of age.
Arm/Group | PR5I (V1) | Pediacel® (V2) | PR5I (V3)
Number analyzed (Participants) | 384 | 383 | 383
Percentage of Participants | 4.9 | 6.3 | 4.7

13. Secondary Outcome: Number of Participants Experiencing a Solicited Injection Site Reaction (ISR) Related to the PR5I/Pediacel® Vaccination
Description: The number of participants experiencing solicited ISRs related to the PRI5 or Pediacel® vaccination was assessed. Solicited ISRs (erythema, pain and swelling) occurring at the PR5I or Pediacel® injection site were always considered related to the PR5I or Pediacel® vaccine, respectively. All AEs/ISRs were recorded on the VRC by the participant's parent(s)/legal representative. Data are presented for the number of participants experiencing solicited ISRs up to Day 5 after each vaccination and after any vaccination.
Time Frame: Up to Day 5 following each vaccination
Population: All participants receiving ≥1 dose of PR5I/Pediacel® vaccination with corresponding safety follow-up data after each vaccination (for V1, V2, and V3 arms) and after any vaccination (for overall V1; V2; V3 arm) with PR5I/Pediacel®.
Measure: Count of Participants; unit: Participants
Arm/Group | PR5I (V1) | Pediacel® (V2) | PR5I (V3) | PR5I (V1); Pediacel® (V2); PR5I (V3)
Number analyzed (Participants) | 385 | 385 | 384 | 385
Participants
  Injection-site erythema | 81 | 65 | 69 | 136
  Injection-site pain | 152 | 97 | 93 | 200
  Injection-site swelling | 68 | 52 | 65 | 121

14. Secondary Outcome: Number of Participants Experiencing a Solicited Injection Site Reaction (ISR) Related to the NeisVac-C® (MCC) Vaccination
Description: The number of participants experiencing solicited ISRs related to the NeisVac-C® (MCC) vaccination was assessed. Solicited ISRs (erythema, pain and swelling) occurring at the NeisVac-C® (MCC) injection site were always considered related to the NeisVac-C® (MCC) vaccine. All AEs/ISRs were recorded on the VRC by the participant's parent(s)/legal representative. Data are presented for the number of participants experiencing solicited ISRs up to Day 5 after each NeisVac-C® vaccination and after any NeisVac-C® vaccination.
Time Frame: Up to Day 5 following each vaccination
Population: All participants receiving ≥1 dose of NeisVac-C® vaccination with corresponding safety follow-up data after each vaccination (for V1 and V2 arms) and after any vaccination (for V1; V2 arm) with NeisVac-C®.
Measure: Count of Participants; unit: Participants
Groups:
- PR5I (V1); Pediacel® (V2): [Vaccination 1]: Single doses of PR5I (V419) + NeisVac-C® + Prevenar 13® by intramuscular (IM) injection + oral RotaTeq®, given at 2 months of age. [Vaccination 2]: Single doses of Pediacel® + NeisVac-C® + Prevenar 13® by IM injection + oral RotaTeq®, given at 4 months of age.
Arm/Group | PR5I (V1) | Pediacel® (V2) | PR5I (V1); Pediacel® (V2)
Number analyzed (Participants) | 385 | 385 | 385
Participants
  Injection-site erythema | 41 | 59 | 85
  Injection-site pain | 113 | 89 | 151
  Injection-site swelling | 34 | 42 | 66

15. Secondary Outcome: Number of Participants Experiencing an Unsolicited Injection Site Reaction (ISR) Related to the PR5I/Pediacel® Vaccination
Description: The number of participants experiencing unsolicited ISRs related to the PRI5 or Pediacel® vaccination was assessed. Unsolicited ISRs occurring at the PR5I or Pediacel® injection site were always considered related to the PR5I or Pediacel® vaccine, respectively. All AEs/ISRs were recorded on the VRC by the participant's parent(s)/legal representative. Data are presented for the number of participants experiencing unsolicited ISRs up to Day 15 after each vaccination and after any vaccination.
Time Frame: Up to Day 15 following each vaccination
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | PR5I (V1) | Pediacel® (V2) | PR5I (V3) | PR5I (V1); Pediacel® (V2); PR5I (V3)
Number analyzed (Participants) | 385 | 385 | 384 | 385
Participants
  Injection-site bruising | 1 | 0 | 0 | 1
  Injection-site discomfort | 0 | 1 | 0 | 1
  Injection-site haematoma | 1 | 1 | 1 | 3
  Injection-site haemorrhage | 0 | 1 | 0 | 1
  Injection-site induration | 5 | 4 | 8 | 16
  Injection-site warmth | 1 | 0 | 1 | 1

16. Secondary Outcome: Number of Participants Experiencing an Unsolicited Injection Site Reaction (ISR) Related to the NeisVac-C® (MCC) Vaccination
Description: The number of participants experiencing unsolicited ISRs related to the NeisVac-C® (MCC) vaccination was assessed. Unsolicited ISRs occurring at the NeisVac-C® (MCC) injection site were always considered related to the NeisVac-C® (MCC) vaccine. All AEs/ISRs were recorded on the VRC by the participant's parent(s)/legal representative. Data are presented for the number of participants experiencing unsolicited ISRs up to Day 15 after each NeisVac-C® vaccination and after any NeisVac-C® vaccination.
Time Frame: Up to Day 15 following each vaccination
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | PR5I (V1) | Pediacel® (V2) | PR5I (V1); Pediacel® (V2)
Number analyzed (Participants) | 385 | 385 | 385
Participants
  Injection-site discolouration | 1 | 0 | 1
  Injection-site haematoma | 0 | 2 | 2
  Injection-site induration | 2 | 2 | 4

17. Secondary Outcome: Number of Participants Experiencing a Solicited Systemic Adverse Event (AE)
Description: The number of participants experiencing solicited systemic AEs (crying, decreased appetite, irritability, somnolence, pyrexia, and vomiting) was assessed. Each day from Day 1 to Day 5 following each vaccination, the participant's parent(s)/legal representative recorded all solicited AEs on the VRC. Data are presented for the number of participants experiencing solicited AEs up to Day 5 after each vaccination and after any vaccination.
Time Frame: Up to Day 5 following each vaccination
Population: All participants receiving ≥1 dose of any vaccination with corresponding safety follow-up data after each vaccination (for V1, V2, and V3 arms) and after any vaccination (for overall V1; V2; V3 arm).
Measure: Count of Participants; unit: Participants
Arm/Group | PR5I (V1) | Pediacel® (V2) | PR5I (V3) | PR5I (V1); Pediacel® (V2); PR5I (V3)
Number analyzed (Participants) | 385 | 385 | 384 | 385
Participants
  Crying | 188 | 131 | 102 | 255
  Decreased appetite | 141 | 88 | 76 | 195
  Irritability | 196 | 154 | 119 | 268
  Pyrexia | 19 | 24 | 18 | 52
  Somnolence | 184 | 126 | 84 | 229
  Vomiting | 56 | 35 | 27 | 88

18. Secondary Outcome: Number of Participants Experiencing an Unsolicited Systemic Adverse Event (AE)
Description: The number of participants experiencing unsolicited systemic AEs was assessed. Data are presented for the number of participants experiencing unsolicited AEs up to Day 15 after each vaccination and after any vaccination.
Time Frame: Up to Day 15 following each vaccination
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | PR5I (V1) | Pediacel® (V2) | PR5I (V3) | PR5I (V1); Pediacel® (V2); PR5I (V3)
Number analyzed (Participants) | 385 | 385 | 384 | 385
Participants | 58 | 53 | 89 | 163

19. Secondary Outcome: Number of Participants Experiencing a Serious Adverse Event (SAE)
Description: An SAE is an adverse event (AE) that: results in death; is life threatening; results in persistent or significant disability or incapacity; results in or prolongs a hospitalization; is a congenital anomaly or birth defect; is a cancer; or may jeopardize the participant, potentially require medical or surgical intervention.
Time Frame: Up to ~6 months (at any time during the study)
Population: All participants receiving ≥1 dose of study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | PR5I (V1); Pediacel® (V2); PR5I (V3)
Number analyzed (Participants) | 385
Participants | 12

ADVERSE EVENTS:
Time Frame: Up to ~6 months (Serious adverse events and deaths were collected for the duration of the study. Solicited ISRs / AEs were collected up to 5 days following each vaccination; unsolicited ISRs / AEs were collected up to 15 days following each vaccination.)
Description: Analysis population includes all participants receiving ≥1 dose of study vaccination.
Arm/Group | PR5I (V1); Pediacel® (V2); PR5I (V3)
All-Cause Mortality (participants affected / at risk) | 0/385
Serious Adverse Events (participants affected / at risk) | 12/385
Other Adverse Events (participants affected / at risk) | 360/385
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PR5I (V1); Pediacel® (V2); PR5I (V3) (N=385)
Bronchiolitis (Infections and infestations) | 5 (5)
Periorbital cellulitis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PR5I (V1); Pediacel® (V2); PR5I (V3) (N=385)
Constipation (Gastrointestinal disorders) | 11 (12)
Diarrhoea (Gastrointestinal disorders) | 15 (17)
Vomiting (Gastrointestinal disorders) | 93 (136)
Crying (General disorders) | 255 (452)
Injection site erythema (General disorders) | 152 (316)
Injection site induration (General disorders) | 19 (21)
Injection site pain (General disorders) | 208 (544)
Injection site swelling (General disorders) | 130 (261)
Pyrexia (General disorders) | 56 (69)
Bronchiolitis (Infections and infestations) | 16 (16)
Conjunctivitis (Infections and infestations) | 11 (11)
Nasopharyngitis (Infections and infestations) | 21 (23)
Respiratory tract infection (Infections and infestations) | 12 (13)
Upper respiratory tract infection (Infections and infestations) | 8 (9)
Decreased appetite (Metabolism and nutrition disorders) | 196 (319)
Somnolence (Nervous system disorders) | 229 (414)
Irritability (Psychiatric disorders) | 268 (499)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 9 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Subsequent to public disclosure of study results, an investigator and colleagues participating in a multicenter study may publish data collected in their center independently. In such case the Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations based on these study results 60 calendar days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential will be deleted prior to submission.